CLINICAL TRIAL: NCT07193914
Title: Adaptation of the ECCCLORE Program for Patients With Addictive and Traumatic Problems: Feasibility and Acceptability
Brief Title: Adaptation of the ECCCLORE Program for Patients With Addictive and Traumatic Problems
Acronym: PEAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NIMAO/2024-2/LTB01
Record Dates: First submitted 2025-09-18; First posted 2025-09-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: PTSD; Addiction; Substance Use Disorders; CBT
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Behavior, Addictive; Substance-Related Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with addiction and trauma issues (Experimental)
  Interventions: Other: ECCCLORE program

INTERVENTIONS:
Other: ECCCLORE program — 2-hour sessions in groups of up to 10 people, once a week for 12 weeks plus 30-minute individual sessions after each group session At the beginning of each session, there will be a discussion about the past week and home practices. This will be followed by an alternation between presentations/explanations of key concepts and associated practices. In the individual sessions the previous session and any difficulties encountered during the group session will be reviewed, as well as to address the implementation of home practices.

SUMMARY:
Complex posttraumatic stress disorder (cPTSD) is characterized by chronic and pervasive disruptions in emotion regulation, identity, and relationships following prolonged or multiple exposures to trauma. It is frequently found in patients with addiction. Individuals with cPTSD have more severe addiction. In addition, the co-occurrence of these two disorders is often associated with certain transdiagnostic processes such as impulsivity. Indeed, PTSD is linked to a higher impulsivity score, which in turn promotes increased substance use. A second process also associated with trauma and addiction is hostile attribution bias.

Thus, the trauma-addiction comorbidity generates multiple behavioral consequences (aggression, increased substance use, etc.) that impact patients' quality of life and represent an important treatment target. Many authors and clinicians have worked on creating treatment programs targeting both disorders, although group format treatment lacks empirical support. Indeed, even though the Seeking Safety program has been shown to be effective in reducing PTSD symptoms and substance use, there is currently no evidence to suggest its superiority.

The ECCCLORE program is a new 6-month cognitive behavioral therapy protocol initially designed for patients with borderline personality disorder, in whom addictive and traumatic issues are common. It is shorter than the standard dialectical behavioral therapy (DBT) program, which focuses on emotional dysregulation, impulsivity, and the traumatic dimension and lasts at least 1 year. It also integrates techniques from other approaches such as Acceptance and Commitment Therapy (ACT), which promotes the acceptance of internal experiences and engagement in actions consistent with values. It notably contains tools for developing emotional, distress tolerance, and interpersonal skills that could adapt to the difficulties generated by trauma and addiction. The objective of this research is to test the feasibility and acceptability of a 12-week ECCCLORE program adapted for patients with addictive and traumatic problems. The study investigators hypothesize that the implementation of this program will demonstrate satisfactory feasibility and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one or more addictions
* ASSIST questionnaire score greater than or equal to 11 for alcohol consumption and greater than or equal to 4 for other substances.
* Diagnosis of PTSD and/or CPTSD assessed using the ITQ scale.
* Ability to understand, write, and read French
* The patient must have given their free and informed consent
* The patient must be a member or beneficiary of a health insurance plan

Exclusion Criteria:

* The subject is participating in an interventional study involving a drug or medical device or a Category 1 study within 3 months prior to inclusion
* The patient is under safeguard of justice or state guardianship
* Patients with a psychotic disorder
* Patients with severe cognitive impairment (MoCA < 10)
* Patients experiencing a manic or hypomanic episode
* Patients experiencing a major depressive episode
* Patients participating in an interventional study involving a drug or medical device or a Category 1 RIPH within 3 months prior to inclusion
* Pregnant, parturient, or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a shortened 12-week ECCCLORE program for patients with addiction and trauma issues | Week 12
  Percentage of participants who attended 8 or more sessions
Dropout rate of a shortened 12-week ECCCLORE program for patients with addiction and trauma issues. | Week 12
  Percentage of participants missing 5 or more sessions
Acceptability of the home practice section of the ECCCLORE program | Week 12
  Percentage of participants completing the exercises 8 or more times out of 12 sessions

SECONDARY OUTCOMES:
Patient-reported trauma | Baseline
  International Trauma Questionnaire (ITQ), where PTSD requires the presence of at least one symptom in each of the three symptom clusters plus at least one indicator of functional impairment corresponding to a score ≥ 2 on one item. CPTSD further requires confirmation of at least one symptom in each cluster of disturbance in self-organization and associated functional impairment.
Patient-reported trauma | Week 12
  International Trauma Questionnaire (ITQ), where PTSD requires the presence of at least one symptom in each of the three symptom clusters plus at least one indicator of functional impairment corresponding to a score ≥ 2 on one item. CPTSD further requires confirmation of at least one symptom in each cluster of disturbance in self-organization and associated functional impairment.
Patient-reported trauma | Week 24
  International Trauma Questionnaire (ITQ), where PTSD requires the presence of at least one symptom in each of the three symptom clusters plus at least one indicator of functional impairment corresponding to a score ≥ 2 on one item. CPTSD further requires confirmation of at least one symptom in each cluster of disturbance in self-organization and associated functional impairment.
Patient-reported addiction | Baseline
  Alcohol, Smoking and Substance Involvement Screening Test (ASSIST), for alcohol a score 0-10 is classed as low risk, 11-26: moderate risk, 27 or more: high risk and for other substances: 0-3: low risk, 4-26: moderate risk, 27 or more: high risk.
Patient-reported addiction | Week 12
  Alcohol, Smoking and Substance Involvement Screening Test (ASSIST), for alcohol a score 0-10 is classed as low risk, 11-26: moderate risk, 27 or more: high risk and for other substances: 0-3: low risk, 4-26: moderate risk, 27 or more: high risk.
Patient-reported addiction | Week 24
  Alcohol, Smoking and Substance Involvement Screening Test (ASSIST), for alcohol a score 0-10 is classed as low risk, 11-26: moderate risk, 27 or more: high risk and for other substances: 0-3: low risk, 4-26: moderate risk, 27 or more: high risk.
Patient-reported impulsivity | Baseline
  UPPS-P questionnaire used to measure positive urgency, negative urgency, lack of premeditation, lack of perseverance and sensation seeking
Patient-reported impulsivity | Week 12
  UPPS-P questionnaire used to measure positive urgency, negative urgency, lack of premeditation, lack of perseverance and sensation seeking
Patient-reported impulsivity | Week 24
  UPPS-P questionnaire used to measure positive urgency, negative urgency, lack of premeditation, lack of perseverance and sensation seeking
Hostile Attribution Bias | Baseline
  Word Sentence Association Paradigm-Hostility (WSAP-H), in which hostile attribution biases are calculated by averaging the scores across the 16 trials with a hostile word. The higher the score, the greater the hostile attribution bias.
Hostile Attribution Bias | Week 12
  Word Sentence Association Paradigm-Hostility (WSAP-H), in which hostile attribution biases are calculated by averaging the scores across the 16 trials with a hostile word. The higher the score, the greater the hostile attribution bias.
Hostile Attribution Bias | Week 24
  Word Sentence Association Paradigm-Hostility (WSAP-H), in which hostile attribution biases are calculated by averaging the scores across the 16 trials with a hostile word. The higher the score, the greater the hostile attribution bias.
Patient-reported aggressivity | Baseline
  Aggression Questionnaire (AQ-12). Items are rated using a 6-point Likert-type scale ranging from 1 "does not apply to me at all" to 6 "applies to me completely".
Patient-reported aggressivity | Week 12
  Aggression Questionnaire (AQ-12). Items are rated using a 6-point Likert-type scale ranging from 1 "does not apply to me at all" to 6 "applies to me completely".
Patient-reported aggressivity | Week 24
  Aggression Questionnaire (AQ-12). Items are rated using a 6-point Likert-type scale ranging from 1 "does not apply to me at all" to 6 "applies to me completely".
Patient-reported flexibility | Baseline
  Multidimensional Psychological Flexibility Inventory Short-Form (MPFI-24), only items 1 to 12 will be tested: acceptance, awareness of the present moment, defusion, self as context, contact with values, and committed actions.
Patient-reported flexibility | Week 12
  Multidimensional Psychological Flexibility Inventory Short-Form (MPFI-24), only items 1 to 12 will be tested: acceptance, awareness of the present moment, defusion, self as context, contact with values, and committed actions.
Patient-reported flexibility | Week 24
  Multidimensional Psychological Flexibility Inventory Short-Form (MPFI-24), only items 1 to 12 will be tested: acceptance, awareness of the present moment, defusion, self as context, contact with values, and committed actions.
Patient-reported depression | Baseline
  Beck Depression Inventory (BDI-21)
Patient-reported depression | Week 12
  Beck Depression Inventory (BDI-21)
Patient-reported depression | Week 24
  Beck Depression Inventory (BDI-21)

CONTACTS AND LOCATIONS:
Overall Officials: Laure Thebault, Principal Investigator — CHU de Nimes
Locations (1):
- CHU de Nîmes, Nîmes, Nîmes, France